CLINICAL TRIAL: NCT02801786
Title: Randomized Study of the Use of Tamoxifen Versus Ointment Lidocaine for Reducing the Pain and Discomfort in Mammography
Brief Title: TAmoxifen Versus LIdocaine Cream. A Randomized Clinical Trial for Reducing Pain and Discomfort During Mammography
Acronym: TALI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Goias (Other)
Responsible Party: Principal Investigator, Ruffo Freitas-Junior, Responsible Party was entered in the old format as Ruffo Freitas-Junior,Federal University of Goias., Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TALI TRIAL
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Pain; Discomfort
Keywords: Mammography; Premedication; Pain; Discomfort; Breast
MeSH Terms: conditions — Pain | interventions — Starch; Lidocaine; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Five capsules containing placebo
  Interventions: Drug: Placebo
- Tamoxifen (Experimental): Five capsules containing 20mg of tamoxifen.
  Interventions: Drug: Placebo; Drug: Tamoxifen
- Lidocaine (Experimental): One sachet containing lidocaine gel at 4%
  Interventions: Drug: Placebo; Drug: Lidocaine

INTERVENTIONS:
Drug: Placebo — The arm will be composed of 03 women who used placebo capsules and gel.
  Other Names: Starch
Drug: Lidocaine — The arm 2 will consist of women who used the placebo capsules for 5 days and 4% lidocaine gel 15 minutes before the test.
  Arms: Lidocaine
Drug: Tamoxifen — The arm 01 is composed of patients who use tamoxifen 20mg one capsule per day for 05 days before the test and placebo gel 15 minutes before the exam.
  Arms: Tamoxifen

SUMMARY:
This is a double-blind placebo-controlled randomized clinical trial to test the use of tamoxifen or lidocaine for diminishing the pain and discomfort while performing mammography, intending to include 450 patients distributed between the three groups.

DETAILED DESCRIPTION:
This is a double-blind placebo-controlled randomized clinical trial to test the use of tamoxifen or lidocaine for diminishing the pain and discomfort while performing mammography, intending to include 450 patients distributed between the three groups.

Inclusion criteria:Patients presenting mastalgia with a prior indication for mammography who is over 40 years old, undergoing their radiological examination at the university hospital of the Federal University of Goias. The only patients who were not included were those who did not wish to participate in the study.

The patients will receive:

* Group 1:Five capsules containing 20mg of tamoxifen plus one sachet containing gel placebo;
* Group 2: Five capsules containing placebo and one sachet containing lidocaine gel at 4%;
* Group 3: Five capsules containing placebo plus one sachet containing gel placebo.

Mammography procedures: The mammography at the university hospital was carried out using a high-resolution mammograph with mean compression in each plane of approximately 800 newtons.

All the patients will undergo at least four imaging views: one craniocaudal and one mediolateral oblique plane for each breast. When necessary, complementary imaging will be used, including selective compression, magnification or other methods.

Control variables:

* Patient's age in completed years at the time of the study;
* Time within the menstrual cycle;
* Menopausal status;
* Use of oral contraceptives;
* Use of hormone replacement therapy;
* Previous history of mastalgia;
* Number of cups of coffee drunk per day;
* Bra size;
* Weight and height, for body mass index (BMI): weight in kilograms and height in meters, according to information provided by the patient at the time of the study;
* Any previous mammographic examination.

Dependent variables:

The pain will be used to measure according to the linear visual analog pain scale. Discomfort will be recorded into four possible categories according to the patient's opinion: no discomfort, uncomfortable, very uncomfortable or intolerable.

Ethical matters:

This study was approved by the Research Ethics Committee of the university hospital of the Federal University of Goias and it will be conducted in accordance with the ruling principles of the Helsinki Convention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mastalgia in the mastology program with age 40 who have indication for mammography.

Exclusion Criteria:

* Patients who do not wish to participate in the study
* Patients who underwent prosthetic silicone implants
* Patients who mammoplasty (breast reduction or mastopexy) were submitted
* Pregnant women
* Patients allergic to tamoxifen or to lidocaine, heart disease, or patients with a history deep vein thrombosis.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Tamoxifen for pain during mammography | Between review, test, randomization, application of results, data analysis and delivery of results for publication will be 24 months.
  An additional 15% of patients who did not experience pain during mammography using the medication.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Goias, Goiânia, Goiás, Brazil

REFERENCES:
- [Result] Kashikar-Zuck S, Keefe FJ, Kornguth P, Beaupre P, Holzberg A, Delong D. Pain coping and the pain experience during mammography: a preliminary study. Pain. 1997 Nov;73(2):165-172. doi: 10.1016/S0304-3959(97)00114-0. PMID 9415502